CLINICAL TRIAL: NCT04481880
Title: Correlation of Intra-abdominal Pressure With Gastric and Urinary Bladder Pressures in Patients With Morbid Obesity
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, rambam75, Dr. Shadi Hamoud, Deputy director, Internal medicine E, Rambam Health Care Campus
Other Study IDs: Rambam ethics number: 0019-12
Record Dates: First submitted 2020-03-22; First posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Morbid Obesity; Intra-Abdominal Hypertension; Bariatric Surgery Candidate
MeSH Terms: conditions — Obesity, Morbid; Intra-Abdominal Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: measuring IAP and respiratory parameters — Effect of IAP on respiratory parameters Correlation between IAP and Gastric and urinary bladder pressures

SUMMARY:
The correlations between gastric and urinary bladder pressures with Intra-abdominal pewssure have not been addressed

DETAILED DESCRIPTION:
Intra-abdominal pressure (IAP) affects cardio-respiratory hemodynamics and can be assessed either directly, or by measuring gastric or urinary bladder pressure. However, in patients with morbid obesity, the correlations between gastric and urinary bladder pressures with IAP have not been addressed. The investigator's aim was to assess the correlations between IAP and gastric and urinary bladder pressure in patients with morbid obesity, at normal and elevated levels of IAP, and to examine the effects of increasing IAP and patient position on hemodynamic and respiratory parameters.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* Morbid Obesity
* candidate for bariatric surgery

Exclusion Criteria:

* Contraindication to laparoscopy
* Advanced COPD
* Advanced CHF

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adult subjects with morbid obesity
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
correlation between intra-abdominal pressure and gastric pressure | Early post-operative- up to 1 week post operation
  different measurement methods
Intra-abdominal pressure | 0-7 days post bariatric surgery
  Correlation between measured IAP according to different measurement methods

IPD SHARING:
Plan to Share IPD: Undecided